CLINICAL TRIAL: NCT04590235
Title: A Phase 1 Open Label Study to Assess the Safety, Tolerability, Pharmacokinetics and Clinical Efficacy of Selumetinib, a Selective Mitogen Activated Protein Kinase Kinase (MEK) 1 Inhibitor, in Chinese Paediatric and Adult Subjects With Neurofibromatosis Type 1 (NF1) and Inoperable Plexiform Neurofibromas (PN)
Brief Title: A Study of Selumetinib in Chinese Paediatric and Adult Subjects With Neurofibromatosis Type 1 (NF1) and Inoperable Plexiform Neurofibromas (PN)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1346C00011
Record Dates: First submitted 2020-07-28; First posted 2020-10-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Neurofibromatosis 1; Neurofibroma Plexiform
Keywords: Neurofibromatosis Type 1; Plexiform Neurofibromas; Phase 1; Selumetinib; Chinese; Paediatric; Adult
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform | interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Selumetinib (Experimental): All eligible subjects will first receive a single oral dose of selumetinib 25 mg/m^2. Then, selumetinib 25 mg/m^2 oral twice daily will be administered continuously until disease progression or unacceptable drug-related toxicity, whichever occurs first.
  Interventions: Drug: Selumetinib

INTERVENTIONS:
Drug: Selumetinib — All eligible subjects will first receive a single oral dose of selumetinib 25 mg/m^2. After a washout period of 2 days, oral selumetinib 25 mg/m^2 twice daily will be administered continuously. Subjects will continue to receive selumetinib until disease progression or unacceptable drug-related toxicity, whichever occurs first.
  10 mg and 25 mg capsules strengths available.
  Other Names: Koselugo

SUMMARY:
A Phase 1 Open Label Study to Assess the Safety, Tolerability, Pharmacokinetics and Clinical Efficacy of Selumetinib, a Selective Mitogen Activated Protein Kinase Kinase (MEK) 1 Inhibitor, in Chinese Paediatric and Adult Subjects with Neurofibromatosis Type 1 (NF1) and Inoperable Plexiform Neurofibromas (PN).

DETAILED DESCRIPTION:
Paediatric and adult patients with Neurofibromatosis Type 1 (NF1) and Inoperable Plexiform Neurofibromas (PN) will be evaluated in the screening visit to confirm eligibility. Approximately 16 paediatric and 16 adult qualified patients will receive oral selumetinib 25 mg/m^2 twice a day (approximately every 12 hours) continuously until disease progression or unacceptable drug-related toxicity, whichever occurs first. Once a patient has discontinued the study treatment then the patient will be followed for specified period for safety assessment

ELIGIBILITY:
Inclusion Criteria:

* Paediatric cohort: Chinese subjects ≥3 years and <18 years of age
* Adult cohort: Chinese subjects ≥18 years of age at the time of study enrollment
* Subjects must be diagnosed with (i) NF1 as per NIH Consensus Development Conference Statement and（ii) PN is defined as a neurofibroma that has grown along the length of a nerve and may involve multiple fascicles and branches. (iii) inoperable PN
* Subjects must have at least one measurable typical or nodular PN
* Absolute neutrophil count ≥1.5×10^9/L, haemoglobin ≥9g/dL, and platelet count ≥100×10^9/L. Subject must be without growth factor support and platelet transfusion support 7 days before the screening assessment.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2×upper limit of normal (ULN), total bilirubin ≤1.5×ULN except in the case of subjects with documented Gilbert's disease (≤2.5×ULN).

Exclusion Criteria:

* Evidence of malignant peripheral nerve sheath tumour.
* Clinically significant cardiovascular disease
* Prior malignancy (except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject had been disease free for ≥2 years or which would not have limited survival to <2 years) or other cancer requiring treatment with chemotherapy or radiation therapy.
* Subjects with the following ophthalmological findings/conditions:

Current or past history of retinal pigment epithelial detachment/central serous retinopathy or retinal vein occlusion; Intraocular pressure >21 mmHg (or ULN adjusted by age) or uncontrolled glaucoma (irrespective of IOP); Subjects with known glaucoma and increased IOP who do not have meaningful vision (light perception only or no light perception) and are not experiencing pain related to the glaucoma, may be eligible after discussion with the study physician; Any other significant abnormality on ophthalmic examination that would make the subject unsuitable for enrolment into the study, as assessed by the investigator.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | For paediatric cohort: from signing the informed consent form until up to 3 years after last subject dosed; For adult cohort: from signing the informed consent form until up to 2 years+30 days after last subject dosed.
  * Occurrence/frequency.
  * Relationship to IP as assessed by investigator.
  * Common Terminology Criteria for Adverse Events (CTCAE) grade.
  * Seriousness.
  * Death.
  * Adverse events leading to discontinuation of IP.
  * Adverse events of special interest.
Area under the concentration-time curve from zero to the last measurable concentration (AUC0-t) of selumetinib and its metabolite (N-desmethyl selumetinib) in Chinese paediatric and adult subjects with NF 1 and inoperable Plexiform Neurofibromas | From the first consent patient first dose to last patient steady state PK collection. Expected duration is approximately 1 year.
  AUC0-t after single dose and multiple doses administration
Maximum plasma concentration (Cmax) of selumetinib and its metabolite (N-desmethyl selumetinib) in Chinese paediatric and adult subjects with NF 1 and inoperable Plexiform Neurofibromas | From the first consent patient first dose to last patient steady state PK collection. Expected duration is approximately 1 year.
  Cmax after single dose and multiple doses administration
Terminal half-life (t1/2) of selumetinib and its metabolite (N-desmethyl selumetinib) in Chinese paediatric and adult subjects with NF 1 and inoperable Plexiform Neurofibromas | From the first consent patient first dose to last patient steady state PK collection. Expected duration is approximately 1 year.
  t1/2 after single dose and multiple doses administration

SECONDARY OUTCOMES:
objective response rate (ORR) of selumetinib in Chinese paediatric and adult subjects with Neurofibromatosis Type 1 and inoperable Plexiform Neurofibromas | First patient first dose until up to 2 years after last subject dosed
  measured by 3D volumetric magnetic resonance imaging (MRI) of the target and nontarget PN
duration of response (DoR) of selumetinib in Chinese paediatric and adult subjects with Neurofibromatosis Type 1 and inoperable Plexiform Neurofibromas | First patient first dose until up to 2 years after last subject dosed
  measured by 3D volumetric magnetic resonance imaging (MRI) of the target and nontarget PN
progression-free survival (PFS) of selumetinib in Chinese paediatric and adult subjects with Neurofibromatosis Type 1 and inoperable Plexiform Neurofibromas | First patient first dose until up to 2 years after last subject dosed
  measured by 3D volumetric magnetic resonance imaging (MRI) of the target and nontarget PN
time to progression (TTP) of selumetinib in Chinese paediatric and adult subjects with Neurofibromatosis Type 1 and inoperable Plexiform Neurofibromas | First patient first dose until up to 2 years after last subject dosed
  measured by 3D volumetric magnetic resonance imaging (MRI) of the target and nontarget PN
time to response (TTR) of selumetinib in Chinese paediatric and adult subjects with Neurofibromatosis Type 1 and inoperable Plexiform Neurofibromas | First patient first dose until up to 2 years after last subject dosed
  measured by 3D volumetric magnetic resonance imaging (MRI) of the target and nontarget PN
Measures of Physical function via Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire | First patient first dose until up to 2 years after last subject dosed
Measures health-related quality of life (HRQoL) via PedsQL (paediatric cohort, self-and parent-reported) | First patient first dose until up to 2 years after last subject dosed
Measures of pain via FLACC scale | First patient first dose until up to 2 years after last subject dosed
Measures health-related quality of life (HRQoL) via EORTC QLQ-C30 (adult cohort) | First patient first dose until up to 2 years after last subject dosed
Measures health-related quality of life (HRQoL) via PlexiQoL (adult cohort) | First patient first dose until up to 2 years after last subject dosed
Measures of pain via Faces Pain Scale (revised) | First patient first dose until up to 2 years after last subject dosed
Measures of pain via NRS-11 | First patient first dose until up to 2 years after last subject dosed
Measures of pain via PII | First patient first dose until up to 2 years after last subject dosed
Measures of pain via Pain Medication Survey | First patient first dose until up to 2 years after last subject dosed

CONTACTS AND LOCATIONS:
Overall Officials: Qingfeng Li, Principal Investigator — Shanghai Ninth People's Hospital affiliated to Shanghai JiaoTong University
Locations (1):
- Research Site, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Clinical Study Protocol Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1346C00011&attachmentIdentifier=556c5830-09c2-4ffb-944a-7f9bcbb2f1e7&fileName=Clinical_Study_Protocol_redacted.pdf&versionIdentifier=
- See also: SAP Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1346C00011&attachmentIdentifier=cde424b4-f974-4e7b-a832-c1e33fe92bf0&fileName=Statistical_Analysis_Plan_redacted.pdf&versionIdentifier=
- See also: CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1346C00011&attachmentIdentifier=f9183afc-3cc5-48d8-aee8-3a8790903b31&fileName=CSR_synopsis_redacted.pdf&versionIdentifier=
- See also: Study Results — https://astrazenecaclinicaltrials.com/study/D1346C00011/